CLINICAL TRIAL: NCT00144612
Title: An Open-label, Extension, Phase III Study to Evaluate the Long-term Safety and Efficacy of MRA in Patients With sJIA Who Participated in Studies MRA011JP or MRA316JP
Brief Title: Long-term Treatment Study of MRA for Systemic Juvenile Idiopathic Arthritis (sJIA)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chugai Pharmaceutical (Industry)
Responsible Party: Chugai Pharmaceutical, Chugai Pharmaceutical
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MRA317JP
Record Dates: First submitted 2005-09-02; First posted 2005-09-05 (Estimated); Last update posted 2009-12-23 (Estimated); Status verified 2009-12

CONDITIONS: Systemic Juvenile Idiopathic Arthritis
MeSH Terms: conditions — Arthritis, Juvenile | interventions — tocilizumab

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: MRA(Tocilizumab)

INTERVENTIONS:
Drug: MRA(Tocilizumab) — 8mg/kg/2weeks

SUMMARY:
An open-label, extension, Phase III study to evaluate the long-term safety and efficacy of MRA in patients with sJIA who were participated in Studies MRA011JP or MRA316JP

ELIGIBILITY:
Inclusion criteria (MRA011JP patients)

* Of the patients who received the three infusions of MRA at the same dose in the main evaluation period in the previous study and are currently in the continued treatment period
* the patients in whom it is confirmed that the drug is effective and there are no problems with safety (MRA316JP patients)
* Patients who proceed to the blind period and in whom the last observations are done after study completion or withdrawal
* Patients who receive the three infusions in the open-label period and do not meet the criteria for transition to the blind period

Exclusion criteria

* Patients who were not enrolled by 3 months after completion of the previous study
* Patients who have been treated with infliximab or etanercept from completion of the previous study until the start of treatment in this study

Ages: 2 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2004-07; Primary Completion 2005-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Efficacy:Percentage of patients showing 30% improvement in the JIA core set compared with before the first infusion of the investigational product (including the previous study) | whole period
Safety:Incidence and severity of adverse events and adverse reactions | whole period
Pharmacokinetics:The time profile of the trough serum MRA concentration at 0W, then every 2Wks | 0 week and every 2 weeks

SECONDARY OUTCOMES:
Efficacy:Time profiles of CRP and ESR, percentage of patients showing 30%, 50%, and 70% improvement in the JIA core set, JIA core set variables, pain, corticosteroid dose at 0W, then every 2Wks | 0 week and every 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Takahiro Kakehi, Study Director — Chugai Pharmaceutical

REFERENCES:
- [Derived] Aoki C, Inaba Y, Choe H, Kaneko U, Hara R, Miyamae T, Imagawa T, Mori M, Oba MS, Yokota S, Saito T. Discrepancy between clinical and radiological responses to tocilizumab treatment in patients with systemic-onset juvenile idiopathic arthritis. J Rheumatol. 2014 Jun;41(6):1171-7. doi: 10.3899/jrheum.130924. Epub 2014 May 1. PMID 24786929
- [Derived] Yokota S, Imagawa T, Mori M, Miyamae T, Takei S, Iwata N, Umebayashi H, Murata T, Miyoshi M, Tomiita M, Nishimoto N, Kishimoto T. Longterm safety and effectiveness of the anti-interleukin 6 receptor monoclonal antibody tocilizumab in patients with systemic juvenile idiopathic arthritis in Japan. J Rheumatol. 2014 Apr;41(4):759-67. doi: 10.3899/jrheum.130690. Epub 2014 Mar 15. PMID 24634205
- [Derived] Yokota S, Imagawa T, Mori M, Miyamae T, Aihara Y, Takei S, Iwata N, Umebayashi H, Murata T, Miyoshi M, Tomiita M, Nishimoto N, Kishimoto T. Efficacy and safety of tocilizumab in patients with systemic-onset juvenile idiopathic arthritis: a randomised, double-blind, placebo-controlled, withdrawal phase III trial. Lancet. 2008 Mar 22;371(9617):998-1006. doi: 10.1016/S0140-6736(08)60454-7. PMID 18358927